CLINICAL TRIAL: NCT05297448
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Assess the Efficacy and Safety of Rifaximin Soluble Solid Dispersion (SSD) for the Delay of Encephalopathy Decompensation in Cirrhosis
Brief Title: Evaluation of Rifaximin SSD for Delaying Encephalopathy Decompensation in Patients With Cirrhosis
Acronym: RED-C-3132
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RNLC3132
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rifaximin SSD-40mg IR (Experimental)
  Interventions: Drug: Rifaximin SSD
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin SSD — Rifaximin Solid Soluble Dispersion Immediate Release Twice Daily
  Arms: Rifaximin SSD-40mg IR
Drug: Placebo — Placebo Twice Daily
  Arms: Placebo

SUMMARY:
Study RNLC3132 is a Phase 3, randomized, double-blind, placebo-controlled, multicenter study to assess the efficacy and safety of rifaximin SSD-40mg IR for the delay of the first episode of overt hepatic encephalopathy (OHE) decompensation in liver cirrhosis, defined by the presence of medically controlled ascites.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of liver cirrhosis with medically controlled ascites (>30 days) not requiring therapeutic paracentesis (could have had paracentesis in the past).
* Conn (West Haven Criteria) score of < 2.
* Mini-Mental State Examination (MMSE) score > 24 at screening.
* ≥ 18 and ≤ 85 years of age.

Key Exclusion Criteria:

* Active COVID-19 that is unresolved
* History of SBP
* History of EVB or AKI-HRS within 6 months
* History of OHE episode (Conn score ≥ 2)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Time to first event of overt hepatic encephalopathy requiring medical intervention in hospital/ER/ED/clinic or death. | 72 weeks

SECONDARY OUTCOMES:
Time to first Conn score ≥ 2 or confirmed OHE requiring medical intervention in hospital/ER/ED/clinic or death | 72 weeks
Time to all-cause hospitalization | 72 weeks
Time to first event of OHE that requires hospitalization, or all-cause death | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mader, Study Director — Bausch Health
Locations (187):
- United States (89):
  - Bausch Site 591, Homewood, Alabama
  - Bausch Site 445, Chandler, Arizona
  - Bausch Site 453, Sun City, Arizona
  - Bausch Site 587, Tucson, Arizona
  - Bausch Site 550, Bakersfield, California
  - Bausch Site 415, Coronado, California
  - Bausch Site 585, Covina, California
  - Bausch Site 592, Fresno, California
  - Bausch Site 582, Lancaster, California
  - Bausch Site 590, Long Beach, California
  - Bausch Site 414, Los Angeles, California
  - Bausch Site 405, Orange, California
  - Bausch Site 482, Valencia, California
  - Bausch Site 575, Colorado Springs, Colorado
  - Bausch Site 425, Doral, Florida
  - Bausch Site 449, Hialeah, Florida
  - Bausch Site 558, Hialeah, Florida
  - Bausch Site 418, Hialeah, Florida
  - Bausch Site 468, Hollywood, Florida
  - Bausch Site 495, Miami, Florida
  - Bausch Site 543, Miami, Florida
  - Bausch Site 479, Miami, Florida
  - Bausch Site 428, Miami, Florida
  - Bausch Site 470, Miami, Florida
  - Bausch Site 486, Miami, Florida
  - Bausch Site 552, Miami, Florida
  - Bausch Site 594, Miami, Florida
  - Bausch Site 456, Miami, Florida
  - Bausch Site 458, Miami, Florida
  - Bausch Site 435, Miami, Florida
  - Bausch Site 452, Miami Lakes, Florida
  - Bausch Site 431/443, Ocala, Florida
  - Bausch Site 450, Ocala, Florida
  - Bausch Site 446, Ocoee, Florida
  - Bausch Site 421, Orange City, Florida
  - Bausch Site 596, Orlando, Florida
  - Bausch Site 537, Palmetto Bay, Florida
  - Bausch Site 407, Port Orange, Florida
  - Bausch Site 454, Wellington, Florida
  - Bausch Site 429, Zephyrhills, Florida
  - Bausch Site 577, Macon, Georgia
  - Bausch Site 475, Gurnee, Illinois
  - Bausch Site 588, South Bend, Indiana
  - Bausch Site 466, West Des Moines, Iowa
  - Bausch Site 524, Topeka, Kansas
  - Bausch Site 457, Lafayette, Louisiana
  - Bausch Site 531, Marrero, Louisiana
  - Bausch Site 488, Metairie, Louisiana
  - Bausch Site 413, New Orleans, Louisiana
  - Bausch Site 442, Shreveport, Louisiana
  - Bausch Site 583, Greenbelt, Maryland
  - Bausch Site 463, Flowood, Mississippi
  - Bausch Site 460, Jefferson City, Missouri
  - Bausch Site 598, Florham Park, New Jersey
  - Bausch Site 597, Freehold, New Jersey
  - Bausch Site 411, Sparta, New Jersey
  - Bausch Site 455, Toms River, New Jersey
  - Bausch Site 436, East Syracuse, New York
  - Bausch Site 401, The Bronx, New York
  - Bausch Site 427, Asheville, North Carolina
  - Bausch Site 494, Monroe, North Carolina
  - Bausch Site 422, Smithfield, North Carolina
  - Bausch Site 410, Dayton, Ohio
  - Bausch Site 580, Liberty Township, Ohio
  - Bausch Site 403, Springboro, Ohio
  - Bausch Site 472, Westlake, Ohio
  - Bausch Site 581, Allentown, Pennsylvania
  - Bausch Site 400, Harrisburg, Pennsylvania
  - Bausch Site 576, Philadelphia, Pennsylvania
  - Bausch Site 484, Providence, Rhode Island
  - Bausch Site 599, Columbia, South Carolina
  - Bausch Site 480, Summerville, South Carolina
  - Bausch Site 423, Chattanooga, Tennessee
  - Bausch Site 434, Chattanooga, Tennessee
  - Bausch Site 579, Hermitage, Tennessee
  - Bausch Site 600, Union City, Tennessee
  - Bausch Site 406, Dallas, Texas
  - Bausch Site 519, Denison, Texas
  - Bausch Site 437, Houston, Texas
  - Bausch Site 447, Humble, Texas
  - Bausch Site 448, San Marcos, Texas
  - Bausch Site 409, Waco, Texas
  - Bausch Site 416, Wichita Falls, Texas
  - Bausch Site 402, Burlington, Vermont
  - Bausch Site 559, Norfolk, Virginia
  - Bausch Site 424, Richmond, Virginia
  - Bausch Site 490, Richmond, Virginia
  - Bausch Site 595, Richmond, Virginia
  - Bausch Site 404, Roanoke, Virginia
- Australia (2):
  - Bausch Site 709, Camperdown, New South Wales
  - Bausch Site 710, Westmead, New South Wales
- Belgium (6):
  - Bausch Site 972, Antwerp
  - Bausch Site 978, Genk
  - Bausch Site 973, Ghent
  - Bausch Site 976, Kortrijk
  - Bausch Site 974, Liège
  - Bausch Site 975, Mechelen
- Bulgaria (6):
  - Bausch Site 982, Rousse
  - Bausch Site 969, Sliven
  - Bausch Site 967, Sofia
  - Bausch Site 968, Sofia
  - Bausch Site 984, Sofia
  - Bausch Site 966, Stara Zagora
- Canada (12):
  - Bausch Site Heritage Medical Research Clinic, Calgary, Alberta
  - Bausch Site University of Alberta Hospital, Edmonton, Alberta
  - Bausch Site G.I.R.I. GI Research Institute, Vancouver, British Columbia
  - Bausch Site Barrie GI Associates, Barrie, Ontario
  - Bausch Site Brampton Civic Hospital, Brampton, Ontario
  - Bausch Site McMaster University Medical Centre - Hamilton Health Services, Hamilton, Ontario
  - Bausch Site Albany Medical Clinic, Toronto, Ontario
  - Bausch Site Toronto General Hospital, Toronto, Ontario
  - Bausch Site: Pharmaceutical Integrated Research Corporation, Waterloo, Ontario
  - Bausch Site Clinique Medicale L'Actuel, Montreal, Quebec
  - Bausch Site: CHUM Centre de Recherche, Montreal, Quebec
  - Bausch Site 605, Québec
- France (14):
  - Bausch Site 804, Angers
  - Bausch Site 818, Belfort
  - Bausch Site 810, Besançon
  - Bausch Site 802, Clermont-Ferrand
  - Bausch Site 808, Limoges
  - Bausch Site 805, Lyon
  - Bausch Site 807, Nice
  - Bausch Site 801, Paris
  - Bausch Site 817, Paris
  - Bausch Site 809, Pessac
  - Bausch Site 815, Rennes
  - Bausch Site 803, Toulouse
  - Bausch Site 813, Vandœuvre-lès-Nancy
  - Bausch Site 811, Villejuif
- Bausch Site 737, Berlin, Germany
- Hungary (2):
  - Bausch Site 859, Budapest
  - Bausch Site 856, Debrecen
- India (6):
  - Bausch Site 352, Belagavi
  - Bausch Site 350, Mangaluru
  - Bausch Site 356, Nagpur
  - Bausch Site 354, Nashik
  - Bausch Site 361, Secunderabad
  - Bausch Site 351, Sūrat
- Italy (5):
  - Bausch Site 881, Milan
  - Bausch Site 883, Napoli
  - Bausch Site 884, Novara
  - Bausch Site 882, Palermo
  - Bausch Site 879, Rozzano
- Bausch Site 970, Ulaanbaatar, Mongolia
- New Zealand (3):
  - Bausch Site 779, Christchurch
  - Bausch Site 776, Grafton
  - Bausch Site 778, Hamilton
- Poland (7):
  - Bausch Site 902, Bydgoszcz
  - Bausch Site 904, Katowice
  - Bausch Site 909, Krakow
  - Bausch Site 901, Mysłowice
  - Bausch Site 903, Staszów
  - Bausch Site 908, Wroclaw
  - Bausch Site 906, Wroclaw
- Puerto Rico (2):
  - Bausch Site 440, Guaynabo
  - Bausch Site 589, San Juan
- South Korea (19):
  - Bausch Site 759, Busan
  - Bausch Site 751, Busan
  - Bausch Site 769, Daegu
  - Bausch Site 764, Daegu
  - Bausch Site 763, Daejeon
  - Bausch Site 768, Gangwon-do
  - Bausch Site 758, Goyang-si
  - Bausch Site 765, Gyeonggi-do
  - Bausch Site 754, Gyeongsang
  - Bausch Site 770, Seongnam-si
  - Bausch Site 757, Seoul
  - Bausch Site 766, Seoul
  - Bausch Site 752, Seoul
  - Bausch Site 762, Seoul
  - Bausch Site 760, Seoul
  - Bausch Site 753, Seoul
  - Bausch Site 767, Seoul
  - Bausch Site 755, Seoul
  - Bausch Site 761, Yongin-si
- Spain (7):
  - Bausch Site 931, Barcelona
  - Bausch Site 937, Madrid
  - Bausch Site 928, Málaga
  - Bausch Site 936, Pontevedra
  - Bausch Site 933, Valencia
  - Bausch Site 935, Valencia
  - Bausch Site 927, Zaragoza
- United Kingdom (5):
  - Bausch Site 941, Dundee
  - Bausch Site 947, Hull
  - Bausch Site 946, Liverpool
  - Bausch Site 945, Nottingham
  - Bausch Site 942, Plymouth

IPD SHARING:
Plan to Share IPD: Undecided